CLINICAL TRIAL: NCT06034301
Title: Feasibility of Interventions Impacting Medication Adherence
Brief Title: Pill Bottle vs Reminder App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202306153
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Medication Adherence
Keywords: Occupational Therapy; Medication Management
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Feasibility randomized controlled trial
Who Masked: Participant
Masking Description: The recruitment material and informed consent will make it appear that the effectiveness between an electronic medication cap and a medication adherence app are being compared and that some participants will get the app while others will get the electronic medication bottle. The reality is that all participants will receive an electronic medication bottle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEMS Cap Only (No Intervention): If the participant is randomized to the control group, they will:
  1. receive a brief education session and be handed a flyer about the importance of medication adherence
  2. receive a MEMS cap and be given instructions on how to use it with their blood pressure medication
- Medication Reminder App + MEMS Cap (Active Comparator): Intervention group that will be shown how to use the mobile phone medication reminder app and be given assistance downloading and setting it up on their personal phone.
  Interventions: Device: Medication Reminder App

INTERVENTIONS:
Device: Medication Reminder App — If the participant is randomized to the intervention group, they will:
  1. receive a brief education session and be handed a flyer about the importance of medication adherence.
  2. get training on how to use the medication reminder app and participant will be given a user guide on how to use the app
  3. demonstrate their understanding on an iPad using the teach back method
  4. install and set up the medication reminder app on their phone
  5. receive a MEMS cap and be given instructions on how to use it with their blood pressure medication. Study team members will use a participant ID to log into the MEMS cap application; no identifiable information will be entered.
  Arms: Medication Reminder App + MEMS Cap

SUMMARY:
Current medication adherence interventions are minimally effective, which results in higher rates of morbidity and mortality for 45 million US adults who have hypertension and low adherence. This feasibility randomized controlled trial seeks to understand the efficacy of reminders and monitoring in the form of a mobile phone application vs usual care on medication adherence as well as the feasibility of the intervention and study procedures. This study will compare participants who use a mobile phone app that notifies them when to take their medications (intervention group) to participants who do not get assigned the app (control group) for 30 days. Medication adherence will be monitored using a Medication Event Monitoring System (MEMS) cap. Both groups will also receive the usual care, which will include giving participants a pamphlet about taking their medications. The long-term goal of this work is to improve antihypertensive medication adherence and to decrease morbidity and mortality. The objective of this application is to test the efficacy of the app based reminders and feedback. The hypothesis driving this research is that the intervention will be more effective than the usual care. The specific aims are as follows:

DETAILED DESCRIPTION:
Current medication adherence interventions are minimally effective, which results in higher rates of morbidity and mortality for 45 million US adults who have hypertension and low adherence. This feasibility randomized controlled trial seeks to understand the efficacy of reminders and monitoring in the form of a mobile phone application vs usual care on medication adherence as well as the feasibility of the intervention and study procedures. This study will compare participants who use a mobile phone app that notifies them when to take their medications (intervention group) to participants who do not get assigned the app (control group) for 30 days. Participants will receive an electronic monitoring cap (i.e. a Medication Event Monitoring System (MEMS) cap) to monitor when they take their antihypertensive medications while they are in the study. Both groups will also receive the usual care, which will include giving participants a pamphlet about taking their medications. The long-term goal of this work is to improve antihypertensive medication adherence and to decrease morbidity and mortality. The objective of this application is to test the efficacy of the app based reminders and feedback. The hypothesis driving this research is that the intervention will be more effective than the usual care. The specific aims are as follows:

Aim 1. Compare the efficacy of the app based reminders and feedback with usual care for the primary outcome of medication adherence in 40 adults with hypertension and low adherence.

Aim 2. Conduct a robust process evaluation to guide intervention improvements, dissemination, and implementation in a diverse sample.

The hypothesis will be tested for two specific aims in 40 adults (20 control, 20 intervention) with hypertension and low adherence. For these aims, the study will be conducted as a phase II single-blind, parallel-group, randomized controlled trial with diverse adults with hypertension over 30 days. Participants will answer surveys about their demographics, knowledge about hypertension, and their medication adherence. They will then be randomized and either be given the standard of care or standard of care plus the intervention (app-based reminders and feedback). The intervention includes a brief training session on downloading and using the medication reminder app. Across arms, Participants will track their medication adherence for 30 days using the MEMS cap. After the 30 days, participants will take surveys about their adherence and knowledge about hypertension and have a brief exit interview with a member of the research team to talk about their experience and debrief them about the study.

ELIGIBILITY:
Inclusion Criteria:

* currently be prescribed an antihypertensive medication by their doctor
* have taken antihypertensive medication for the last year
* be willing to download and use a new app on their phone for the study
* score a 34 or lower on the Hill Bone compliance scale

Exclusion Criteria:

* need assistance taking their medications
* have a severe cognitive impairment
* have a severe visual impairment that prevents them from reading notifications on their phone
* use a pillbox to take their medications
* do not use a smart phone or their smart phone does not meet the requirements for the app to be downloaded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Medication Event Monitoring System (MEMS) Cap | 30 days
  The Medication Event Monitoring System (MEMS) measures medication adherence over 30 days at home. In this system, an electronic cap will be placed on a bottle assigned to the participant's antihypertensive medication and records each time the medication bottle is opened. All participants will use the electronic monitoring for one antihypertensive medication taken daily.
Exit interview | 30 days
  In the exit interview, participants will be asked qualitative questions about their experiences in the study and using the MEMS cap and medication reminder app. This will support a robust process evaluation to guide intervention improvements, dissemination, and implementation in a diverse sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Schwartz, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publications, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal.
URL: https://beckerdms.wustl.edu/

REFERENCES:
- [Background] Ahmed I, Ahmad NS, Ali S, Ali S, George A, Saleem Danish H, Uppal E, Soo J, Mobasheri MH, King D, Cox B, Darzi A. Medication Adherence Apps: Review and Content Analysis. JMIR Mhealth Uhealth. 2018 Mar 16;6(3):e62. doi: 10.2196/mhealth.6432. PMID 29549075
- [Background] Aldeer M., Javanmard M., & Martin R. P. (2018). A review of medication adherence monitoring technologies. Applied System Innovation, 1(2), 2. https://doi: 10.3390/asi1020014.
- [Background] Morrissey EC, Casey M, Glynn LG, Walsh JC, Molloy GJ. Smartphone apps for improving medication adherence in hypertension: patients' perspectives. Patient Prefer Adherence. 2018 May 14;12:813-822. doi: 10.2147/PPA.S145647. eCollection 2018. PMID 29785096
- [Background] Santo K, Chow CK, Thiagalingam A, Rogers K, Chalmers J, Redfern J. MEDication reminder APPs to improve medication adherence in Coronary Heart Disease (MedApp-CHD) Study: a randomised controlled trial protocol. BMJ Open. 2017 Oct 8;7(10):e017540. doi: 10.1136/bmjopen-2017-017540. PMID 28993388
- [Background] Santo K, Singleton A, Chow CK, Redfern J. Evaluating Reach, Acceptability, Utility, and Engagement with An App-Based Intervention to Improve Medication Adherence in Patients with Coronary Heart Disease in the MedApp-CHD Study: A Mixed-Methods Evaluation. Med Sci (Basel). 2019 Jun 4;7(6):68. doi: 10.3390/medsci7060068. PMID 31167489
- [Background] Santo K, Singleton A, Rogers K, Thiagalingam A, Chalmers J, Chow CK, Redfern J. Medication reminder applications to improve adherence in coronary heart disease: a randomised clinical trial. Heart. 2019 Feb;105(4):323-329. doi: 10.1136/heartjnl-2018-313479. Epub 2018 Aug 27. PMID 30150326